CLINICAL TRIAL: NCT03865225
Title: Effects of Heart Rate Variability Biofeedback in Patients With Acute Ischaemic Stroke: Protocol for Randomized Controlled Trial
Brief Title: Effects of Heart Rate Variability Biofeedback in Patients With Acute Ischemic Stroke
Acronym: Strokeback01
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: Michael J. Fox Foundation for Parkinson's Research (Other); University Hospital Carl Gustav Carus (Other)
Responsible Party: Principal Investigator, Timo Siepmann, MD, Assistant Professor, Doctor of Medicine, Principal Investigator, Head of neurological emergency room, University Hospital Carl Gustav Carus, University Hospital Carl Gustav Carus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: EK389102018
Record Dates: First submitted 2019-03-03; First posted 2019-03-06 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Acute Ischaemic Stroke; Autonomic Dysfunction
Keywords: Ischaemic Stroke; Heart Rate Variability; Autonomic Nervous System; cardiac autonomic dysfunction; sudomotor function; vasomotor function
MeSH Terms: conditions — Primary Dysautonomias; Ischemic Stroke | interventions — Biofeedback, Psychology

STUDY DESIGN:
Who Masked: Participant
Masking Description: Sham biofeedback intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group acute ischaemic stroke (Sham Comparator): Acute ischaemic stroke patients receiving 9 x 10 minutes sham-biofeedback over a period of three days
  Interventions: Other: Sham-Biofeedback
- Treatment group acute ischaemic stroke (Active Comparator): Acute ischaemic stroke patients receiving 9 x 10 minutes biofeedback sessions over period of three days
  Interventions: Other: Biofeedback

INTERVENTIONS:
Other: Biofeedback — 9 x 10 minutes biofeedback sessions over period of three days
  Arms: Treatment group acute ischaemic stroke
Other: Sham-Biofeedback — 9 x 10 minutes sham-biofeedback sessions over period of three days
  Arms: Control group acute ischaemic stroke

SUMMARY:
This explorative prospective study aims to assess the effects of heart rate variability biofeedback (HRV biofeedback) in patients with acute ischaemic stroke. Furthermore, the investigators aim to examine the impact of the intervention on cardiac autonomic function and further autonomic parameters such as sudomotor (sympathetic perspiratory gland function) and vasomotor function (sympathetic arterial function). Patients testing is going to be conducted at the Department of Neurology, University Hospital Carl Gustave Carus, Dresden, Germany.

DETAILED DESCRIPTION:
Background:

Ischaemic stroke is among the most common causes for severe disability and death in the industrialized world with steadily increasing prevalence due to the demographic change. Thus more than 795,000 people yearly have a stroke in the United States of America, of which circa 610,000 people have new strokes or a stroke for the first time in their life (Benjamin, et al. 2017). Symptoms of ischaemic stroke patients include dysregulation of the autonomic nervous system such as cardiac and vascular autonomic dysfunction, which correlate with increased mortality and poor functional outcome. This study aims to assess the effects of heart rate variability biofeedback (HRV-Biofeedback) in patients with acute ischaemic stroke. Furthermore, the investigators aim to examine the impact of the intervention on cardiac autonomic function and further autonomic parameters such as sudomotor (sympathetic perspiratory gland function) and vasomotor function (sympathetic arterial function).

Methods/design:

An explorative prospective study is undertaken in 48 patients with acute ischaemic stroke who undergo either 9 x 10-minutes lasting biofeedback sessions over a period of 3 days, or sham-biofeedback (control-group) also over a period of 3 days under randomized controlled conditions.

The HRV-biofeedback technique is based on the recording and visualization of heart rate variability, which is visible in real-time for the patient on a computer screen. In the training sessions, the patient is instructed to breath in a predefined frequency, which has been shown to yield optimal neurologic-cardiac regulation (respiratory sinus arrhythmia) with high heart rate variability. Sham-biofeedback takes place under identical testing and environmental conditions with subjects looking at a computer screen but not having heart rate variability recorded and visualized. Moreover, the patients do not follow any breathing instructions, which could possibly have any influence on the heart rate variability. The sham intervention is applied to rule out any placebo effect.

Before the first and after the last biofeedback-session, measurements of heart rate variability and polygraphical recordings of further autonomic functions (sudomotor function and vasomotor function) are undertaken. Severity of the autonomic functions is captured by a specific survey (Survey of Autonomic Symptoms). The modified Rankin Scale is used to assess functional outcome after acute ischaemic stroke at baseline, with the conclusion of the biofeedback-sessions, and in the context of a telephone-interview after a period of 3 months. Furthermore, severity of common stroke related symptoms is recorded at baseline and after the last training session using the National Institutes of Health Stroke Scale. All assessments as well as all biofeedback training sessions take place at the Stroke Unit of the Department of Neurology, University Hospital Carl Gustave Carus Dresden, Germany.

ELIGIBILITY:
Inclusion Criteria:

* male and female subjects aged between 18 and 90
* written and oral informed consent
* evidence of an ischaemic lesion on cranial computed tomography scan or magnetic resonance imaging

Exclusion Criteria:

* intake of any tricyclic antidepressant within the last 14 days
* atrial fibrillation
* prior diagnosed autonomic neuropathy
* malignant cerebral infarct or indication for treatment at intensive care unit
* aphasia or cognitive deficit with resulted inability to participate in Heart rate variability-biofeedback training
* respiratory insufficiency
* blindness, deafness or other physical limitations with resulted inability to participate in heart rate variability-biofeedback training

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2018-11-25 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Heart rate variability in acute ischaemic stroke patients | Change from Baseline Heart rate variability at 3 days
  Measurement of heart rate variability in acute ischaemic stroke patients
Severity of autonomic symptoms | Change from Baseline Severity of autonomic symptoms at 3 days and at 3 months
  Assessment of autonomic symptoms with Survey of Autonomic Symptoms
Measurement of sudomotor and vasomotor function | Change from Baseline Measurement of sudomotor and vasomotor function at 3 days
  Assessment of sudomotor and vasomotor function in patients with acute ischaemic stroke prior and after intervention

SECONDARY OUTCOMES:
Severity of neurological stroke symptoms | Change from Baseline Severity of neurological stroke symptoms at 3 days
  Assessment of severity of neurological symptoms in patients with acute ischaemic stroke with the National Institutes of Health Stroke Scale (range from 0 to 42)
Degree of disability in patients with acute ischemic stroke | Change from Baseline Functional Outcome at 3 days and at 3 months
  Assessment of functional outcome as the degree of disability in patients with acute ischaemic stroke with the modified Rankin Scale (range from 0 to 6)

CONTACTS AND LOCATIONS:
Overall Officials: Timo Siepmann, PD, MD, Principal Investigator — University Hospital Carl Gustav Carus Dresden, Germany
Locations (1):
- Department of Neurology, University Hospital Carl Gustav Carus Dresden, Germany, Dresden, Saxony, Germany

REFERENCES:
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Derived] Siepmann T, Ohle P, Sedghi A, Simon E, Arndt M, Pallesen LP, Ritschel G, Barlinn J, Reichmann H, Puetz V, Barlinn K. Randomized Sham-Controlled Pilot Study of Neurocardiac Function in Patients With Acute Ischaemic Stroke Undergoing Heart Rate Variability Biofeedback. Front Neurol. 2021 May 26;12:669843. doi: 10.3389/fneur.2021.669843. eCollection 2021. PMID 34122314